CLINICAL TRIAL: NCT00413088
Title: Clinical Trial to Assess Bemiparin Pharmacokinetics at Therapeutic (115 IU/kg) and Prophylactic Doses (3500 IU) Administered Subcutaneously in Single or Multiple Doses in Renal Insufficiency and in the Elderly
Brief Title: Study to Assess Bemiparin Pharmacokinetics in Renal Insufficiency and in the Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Medical Deparment, Rovi Pharmaceuticals Laboratories
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROV-BEM-2005-01
Record Dates: First submitted 2006-12-14; First posted 2006-12-19 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-03

CONDITIONS: Renal Insufficiency
Keywords: renal insufficency; low molecular weight heparin; pharmacokinetics; elderly
MeSH Terms: conditions — Renal Insufficiency | interventions — bemiparin

INTERVENTIONS:
Drug: bemiparin

SUMMARY:
Open pharmacokinetic study with 5 parallel groups and two treatment phases (bemiparin 3,500 IU multiple dose and bemiparin 115 IU/kg single dose). The bemiparin pharmacokinetic profile will be assessed by measuring its effects on the coagulation cascade. Plasma anti-Xa activity (measured using chromogenic amidolytic assay) in IU per milliliter will be the primary endpoint to assess the pharmacokinetic profile of bemiparin.

ELIGIBILITY:
Inclusion Criteria:

Non-elderly healthy volunteers (Group I):

* Male or female subjects aged between 18 and 65 years
* body weight, clinical history, physical examination, vital signs (systolic and diastolic blood pressure, heart beat rate and body temperature), ECG and laboratory tests (hemogram and biochemistry) within normal range
* without evidence of significant organic or psychiatric illness
* who have accepted to participate in the study and have signed the written informed consent.

Patients with renal insufficiency (Groups II, III and IV):

* Male or female subjects aged between 18 and 65 years, who will be assigned to one of the following groups according to renal function:

  * Group II: mild renal insufficiency (creatinine clearance > 50 to 80 ml/min);
  * Group III: Moderate renal insufficiency (creatinine clearance: 30 to 50 ml/min);
  * Group IV: Severe renal insufficiency (creatinine clearance < 30 ml/min). The degree of renal insufficiency will be calculated on the basis of determination of creatinine clearance measuring total urinary output over a 24-h period and serum creatinine levels. Urine samples will be collected no more than 2 weeks before the first experimental period.
* Patients with renal insufficiency must have a stable renal function during the 3 months before their inclusion in the study.
* They must have a body weight between 45 and 110 Kg.
* They have to accept to participate in the study and have signed the written informed consent.

Elderly healthy volunteers (Group V):

* Male or female subjects aged > 65 years old who fulfill with the remaining inclusion criteria specified for non-elderly healthy volunteers.

Exclusion Criteria:

Non-elderly healthy volunteers (Group I):

* Previous history of alcoholism or drugs consumption
* Important consumer of exciting drinks
* Hypersensitivity, allergy, idiosyncrasy to medicines
* Taking another medication four weeks before the initiation of the trial including medication without prescription and medicinal plants
* Positive serology of hepatitis B, C or HIV virus
* History or clinic evidence of concomitant disease
* Familiar history of coagulation's disorders
* surgery within the previous 6 months
* Women who are pregnant or who are not using effective contra conceptive methods
* Ethanol, cannabis, cocaine, amphetamine, benzodiazepin or opiate in urine
* Current platelet count < 100.000/mm3 or serum K > 5,5 mEq/L
* Any contraindication to bemiparin administration in order to authorized summary product characteristics
* Healthy volunteers who are not participating in another clinical trial or have not done so in the past 2 months
* To give blood in the four weeks before beginning of the trial

Patients with renal insufficiency or elderly healthy volunteers (Groups II, III, IV, V):

* Previous history of alcoholism or drugs consumption
* Important consumer of exciting drinks
* Hypersensitivity, allergy, idiosyncrasy to medicines
* Treatment with enzymatic inhibitors or inductors medicines
* Administration with ASA of dosis > 125 mg/day and/or NDAIs with half-life > 20 hours or with high antiagregant effect during the previous ten days to the inclusion
* Chronic hepatopatology
* bilirubin levels > 1,5 mg/dl and/or increment of AST/ALT levels twice higher than maximum limit of normality
* prothrombin time 20% higher than maximun limit of normality and haemoglobine < 8gr/dl or albumim levels <3gr/dl
* Previous history of acute infarction of myocardium, cardiac ischemic or arrhythmia
* Acute illness in the previous week to the participation
* Familiar history of coagulation's disorders
* surgery within the previous 6 months
* Women who are pregnant or who are not using effective contra conceptive methods
* Ethanol, cannabis, cocaine, amphetamine, benzodiazepin or opiate in urine
* Current platelet count < 75.000/mm3 or serum K > 6 mEq/L
* Any contraindication to bemiparin administration in order to authorized summary product characteristics
* Healthy volunteers who are not participating in another clinical trial or have not done so in the past 2 months
* To give blood in the four weeks before beginning of the trial
* Subjects in haemodialysis or peritoneal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-03; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics of bemiparin administered subcutaneously once daily for 4 days at prophylactic doses (3500 IU) and at a single therapeutic dose (115 IU/kg), in renal insufficiency and in the elderly.

SECONDARY OUTCOMES:
To assess the safety and tolerability of bemiparin in all volunteers and patients.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Barbanoj, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau and Fundació Puigvert, Barcelona, Barcelona, Spain